CLINICAL TRIAL: NCT03439449
Title: Computerized, Patient-entered Medical Histories for Managing Chest Pain in the Emergency Department
Brief Title: Computerized Medical History Taking for Acute Chest Pain
Acronym: CLEOS-CPDS
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Thomas Kahan, Professor, Karolinska Institutet
Other Study IDs: KI-CLEOS-CPDS
Record Dates: First submitted 2018-02-07; First posted 2018-02-20 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Chest Pain; Acute Coronary Syndrome
Keywords: History taking, Risk stratification
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood samples with markers of cardiovascular risk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CLEOS software program — Computer-assisted history taking program
Procedure: Physician taken history — Conventional history taking by physicians

SUMMARY:
The aim is to determine the additional value of computerized, patient-entered medical histories for the management of patients presenting at the emergency department with chest pain.

DETAILED DESCRIPTION:
The purpose of this study is to determine the value of a detailed medical history, acquired by computer-directed, patient self-entry of data, for efficient disposition of patients presenting to the emergency department (ED) with chest pain and non-diagnostic first ECG and/or serum markers for acute coronary syndrome (ACS). The research questions posed are: will the added data and systems-based analysis of the data provided by computerization of these processes, as compared with routine physician-acquired histories and analysis; (1) safely risk stratify patients with chest pain, and (2) save time and resources?

Computerized, patient-entered histories will be collected with the software program CLEOS running on tablets (iPad®, Apple Inc, Cupertino, California, USA). The histories to be collected include demographic data, present illness, systems review, past medical history, prescription drugs, previous adverse drug reactions, social history, life-style risks, and family history. Histories will be collected during wait times in the ED, e.g., before patients are seen by a physician and while patients wait for reports of laboratory data collected by routine care.

Data acquired by CLEOS will be related to clinical outcomes in the acute setting and at 30 days and 1 year post-presentation for patients without documented ACS in the acute setting. Outcomes for all patients will be extracted from hospital records and national registries.

For the validation and future development of CLEOS, interviews with patients for the evaluation of patient experience regarding feasibility, acceptance, comprehensiveness and technical aspects of answering the CLEOS interview will take place within one to three months after the ED visit.

This is an exploratory study in which the calculation of the number of participating patients is based on the desired precision of sensitivity and specificity. Assuming that the prevalence is 0.5 (50 %), a power calculation with nQuery® version 7.0 (Statistical Solutions Ltd, Boston, Massachusetts, USA) shows that with 1000 patients the estimated precision of sensitivity and specificity is ±0.03 (3 %). The more the extreme the result, i.e. sensitivity or specificity approaching 0 or 1 (100 %), the higher the precision. The models will be developed in the first 50% of the data acquired (training data set) and validated in the last 50% of the data acquired (validation data set). We also intend to make estimates in subgroups. To ascertain that such estimates can be done, an even larger number of patients must be recruited. Thus, the study intends to recruit data from approximately 2000 patients.

Taken together, this study:

1. will evaluate established clinical guidelines risk scores, as populated with CLEOS data, and compare these results with data obtained during the concurrent ED visit and made available in the standard hospital medical records;
2. will assess how data collected with CLEOS in combination with established risk scores can rule-in and rule-out a diagnosis of an ACS, we will calculate sensitivity, specificity and negative and positive predictive value;
3. aim to develop new risk prediction scores for patients with chest pain, based on data collected with CLEOS; and
4. will evaluate economic aspects of routine care, as compared with management by CLEOS by using standard health economy procedures and analyses to determine the resource utilization and cost differences between management according to guidelines, based on data collected with CLEOS, and current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain recorded by a triage nurse or registrar
* Fluency in Swedish or English
* Non-diagnostic first ECG and/or serum markers
* Manchester triage 2-5
* Informed consent

Exclusion Criteria:

* Inability to carry out computerized history-taking on the dedicated device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presenting at the emergency department with chest pain as presenting complaint.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
A correct diagnosis of an acute coronary syndrome by use of computer-assisted patient entered history or standard history obtained by the cardiologist in attendance | 7 days
  The primary objective is to determine whether the use of computer-assisted patient entered history is better than a standard history obtained by the cardiologist in attendance for the prediction and safe exclusion of an acute coronary syndrome (ACS) in the acute setting in patients with non-diagnostic ECG and/or serum markers. Thus, the primary endpoint is the comparison between the two methods for the proportion of patients with a correct diagnosis of ACS or not ACS in the acute setting, The diagnosis of ACS or not ACS is defined as a validated clinical endpoint within 7 days

SECONDARY OUTCOMES:
A correct exclusion of an acute coronary syndrome up to 30 days by use of computer-assisted patient entered history or standard history obtained by the cardiologist in attendance | 30 days
  To determine whether the use of computer-assisted patient entered history is better than a standard history obtained by the cardiologist in attendance to exclude an acute coronary syndrome (ACS) in the acute setting in patients with non-diagnostic ECG and/or serum markers. Thus, this secondary endpoint is the comparison between the two methods for the proportion of patients with a correct exclusion of ACS in the acute setting, The diagnosis of ACS is defined as a validated clinical endpoint within 30 days
A correct exclusion of an acute coronary syndrome up to 1 year by use of computer-assisted patient entered history or standard history obtained by the cardiologist in attendance | 1 year
  To determine whether the use of computer-assisted patient entered history is better than a standard history obtained by the cardiologist in attendance to exclude an acute coronary syndrome (ACS) in the acute setting in patients with non-diagnostic ECG and/or serum markers. Thus, this secondary endpoint is the comparison between the two methods for the proportion of patients with a correct exclusion of ACS in the acute setting, The diagnosis of ACS is defined as a validated clinical endpoint within 1 year
Direct costs for a patient with a diagnosis of an acute coronary syndrome when patient selection is based on computer-assisted patient entered history, as compared to standard history obtained by the cardiologist in attendance | 1 year
  To measure direct costs for a patient with a diagnosis of an acute coronary syndrome when patient selection is based on computer-assisted patient entered history, as compared to standard history obtained by the cardiologist in attendance. Costs will be obtained patient-by-patient from medical records
Patient experience with computer-assisted patient entered history measured as he proportion of patients who complete a computer-assisted patient entered history | 7 days
  To evaluate the proportion of patients who complete a full computer-assisted patient entered history.
The ability of computer-assisted patient entered history, as compared to standard history obtained by the cardiologist in attendance to provide information required to calculate a TIMI risk score for an ACS. | 7 and 30 days
  To compare the proportions of patients with computer-assisted patient entered history, as compared to standard history obtained by the cardiologist in attendance, where there is sufficient information documented to calculate the Thrombolysis In Myocardial Infarction (TIMI) score. The TIMI score contains the following information: Age, risk factors for coronary artery disease (family history, hypertension, hypercholesterolemia, diabetes, current smoker), a significant coronary artery stenosis, ST segment deviation on the ECG, 2 or more anginal attacks within 24 h, use of aspirin within 7 days, and elevated serum cardiac biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kahan, MD, PhD, Study Chair — Karolinska Institutet; Helge Brandberg, MD, Study Director — Karolinska Institutet; Sabine Koch, PhD, Study Director — Karolinska Institutet; Jonas Spaak, MD, PhD, Study Director — Karolinska Institutet; Carl Johan Sundberg, MD, PhD, Study Director — Karolinska Institutet; David Zakim, MD, PhD, Study Director — Karolinska Institutet
Locations (1):
- Danderyd University Hospital Corp., Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brandberg H, Sundberg CJ, Spaak J, Koch S, Kahan T. Are medical history data fit for risk stratification of patients with chest pain in emergency care? Comparing data collected from patients using computerized history taking with data documented by physicians in the electronic health record in the CLEOS-CPDS prospective cohort study. J Am Med Inform Assoc. 2024 Jun 20;31(7):1529-1539. doi: 10.1093/jamia/ocae110. PMID 38781350
- [Result] Sundberg K, Adeli A, Brandberg H, Spaak J, Koch S, Sundberg CJ, Zakim D, Kahan T, Fritzell K. User experience of self-reported computerized medical history taking for acute chest pain: The Clinical Expert Operating System Chest Pain Danderyd Study. Health Expect. 2022 Dec;25(6):3053-3061. doi: 10.1111/hex.13612. Epub 2022 Sep 23. PMID 36148691
- [Derived] Brandberg H, Schierenbeck F, Sundberg CJ, Koch S, Spaak J, Kahan T. Performance of computerized self-reported medical history taking and HEAR score for safe early rule-out of cardiac events in acute chest pain patients: the CLEOS-CPDS prospective cohort study. Eur Heart J Digit Health. 2024 Nov 12;6(1):104-114. doi: 10.1093/ehjdh/ztae087. eCollection 2025 Jan. PMID 39846077
- [Derived] Zakim D, Brandberg H, El Amrani S, Hultgren A, Stathakarou N, Nifakos S, Kahan T, Spaak J, Koch S, Sundberg CJ. Computerized history-taking improves data quality for clinical decision-making-Comparison of EHR and computer-acquired history data in patients with chest pain. PLoS One. 2021 Sep 27;16(9):e0257677. doi: 10.1371/journal.pone.0257677. eCollection 2021. PMID 34570811
- [Derived] Brandberg H, Sundberg CJ, Spaak J, Koch S, Zakim D, Kahan T. Use of Self-Reported Computerized Medical History Taking for Acute Chest Pain in the Emergency Department - the Clinical Expert Operating System Chest Pain Danderyd Study (CLEOS-CPDS): Prospective Cohort Study. J Med Internet Res. 2021 Apr 27;23(4):e25493. doi: 10.2196/25493. PMID 33904821
- [Derived] Brandberg H, Kahan T, Spaak J, Sundberg K, Koch S, Adeli A, Sundberg CJ, Zakim D. A prospective cohort study of self-reported computerised medical history taking for acute chest pain: protocol of the CLEOS-Chest Pain Danderyd Study (CLEOS-CPDS). BMJ Open. 2020 Jan 21;10(1):e031871. doi: 10.1136/bmjopen-2019-031871. PMID 31969363